CLINICAL TRIAL: NCT00374153
Title: Dismantling Motivational Interviewing and Feedback for College Drinkers
Brief Title: Southern Methodist Alcohol Research Trial (SMART)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Scott T. Walters, PhD, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-06-0310; NIAAA, 1 R01 AA016005-01
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Alcohol Consumption
Keywords: Alcohol; Drinking; College; Motivational; Feedback; Assessment
MeSH Terms: conditions — Alcohol Drinking | interventions — Motivational Interviewing

ARMS (5):
- 1 (Experimental): Online personal feedback report.
  Interventions: Behavioral: Feedback
- 2 (Experimental): In-person Motivational Interview with personal feedback report
  Interventions: Behavioral: Motivational Interview with Feedback
- 3 (Experimental): In-person Motivational Interview only (without a personal feedback report)
  Interventions: Behavioral: Motivational Interview
- 4 (No Intervention): Assessment only
- 5 (No Intervention): Delayed Assessment

INTERVENTIONS:
Behavioral: Feedback — Online personal feedback report
  Arms: 1
Behavioral: Motivational Interview with Feedback — In-person Motivational Interview with personal feedback report
  Arms: 2
Behavioral: Motivational Interview — In-person Motivational Interview only (without a personal feedback report)
  Arms: 3

SUMMARY:
The purpose of this study is to look at the effects of assessment, feedback and motivational interviewing on alcohol consumption among college drinkers.

DETAILED DESCRIPTION:
Excessive alcohol consumption has been a growing problem at many US colleges. In response, colleges and universities have instituted a range of alcohol intervention and prevention programs for students. Motivational Interviewing (MI) is one brief intervention that has been shown to reduce heavy drinking among college students. To date, all college studies of MI have used a format that includes an assessment and feedback delivered in an MI style. Although this format has considerable empirical support, it remains unclear which of the components is necessary to produce behavior change. This study will evaluate the separate and collective effects of MI and feedback among "binge" drinking college students. Additionally, this study will evaluate the effects of the initial drinking assessment, through including a delayed-assessment control group. After an initial screen, 350 students at Southern Methodist University who report at least one heavy (i.e., "binge") episode during the previous two weeks will be randomized to: (1) MI with feedback, (2) MI without feedback, (3) Mailed feedback only, (4) Assessment only, or (5) Delayed assessment only. MI sessions will be delivered by trained and supervised counselors. Participants will be assessed via a secure Internet site at baseline, 3, 6 and 12 months (12 months only for the Delayed-assessment group), with primary outcome measures including self-reported quantity and frequency of drinking, and drinking-related problems. Since college drinking is associated with substantial negative effects for drinkers, as well as for others, the findings of this study may have significant public health implications in terms of reducing costs, and improving services for students who choose to drink.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be enrolled in Southern Methodist University.
* Participants must report one "binge" episode (4 or more drinks in one setting for women, 5 or more drinks in one setting for men) in the past two weeks.
* Participants must be at least 18 years old.

Exclusion Criteria:

* Participants will be excluded if they are not enrolled at Southern Methodist University.
* Participants will be excluded if they do not report at least one "binge" episode in the past two weeks.
* Participants will be excluded if they are less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Drinks per week | one year
Peak BAC | one year

SECONDARY OUTCOMES:
Alcohol Related Consequences (RAPI) | one year
Interpersonal Violence (CADRI) | one year
Readiness to Change (RTCQ) | one year
Protective Behaviors (PBQ) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Walters, PhD, Principal Investigator — University of Texas School of Public Health
Locations (2):
- United States (2):
  - Southern Methodist University, Dallas, Texas
  - University of Texas School of Public Health Dallas Regional Campus, Dallas, Texas

REFERENCES:
- [Result] Walters ST, Roudsari BS, Vader AM, Harris TR. Correlates of protective behavior utilization among heavy-drinking college students. Addict Behav. 2007 Nov;32(11):2633-44. doi: 10.1016/j.addbeh.2007.06.022. Epub 2007 Jun 29. PMID 17669596
- [Result] Walters ST, Vader AM, Harris TR, Field CA, Jouriles EN. Dismantling motivational interviewing and feedback for college drinkers: a randomized clinical trial. J Consult Clin Psychol. 2009 Feb;77(1):64-73. doi: 10.1037/a0014472. PMID 19170454
- [Result] Roudsari BS, Leahy MM, Walters ST. Correlates of dating violence among male and female heavy-drinking college students. J Interpers Violence. 2009 Nov;24(11):1892-905. doi: 10.1177/0886260508325492. Epub 2008 Nov 3. PMID 18981192
- [Result] Harris TR, Walters ST, Leahy MM. Readiness to change among a group of heavy-drinking college students: correlates of readiness and a comparison of measures. J Am Coll Health. 2008 Nov-Dec;57(3):325-30. doi: 10.3200/JACH.57.3.325-330. PMID 18980889
- [Derived] Walters ST, Vader AM, Harris TR, Jouriles EN. Reactivity to alcohol assessment measures: an experimental test. Addiction. 2009 Aug;104(8):1305-10. doi: 10.1111/j.1360-0443.2009.02632.x. PMID 19624323